CLINICAL TRIAL: NCT00742248
Title: Double Blind, Double Dummy, Multicentre, Randomised, Placebo- Controlled, Crossover Design Clinical Trial of 12 μg (Single Dose and Repeated Doses) Formoterol Fumarate Administered Via pMDI With HFA-134a Propellant or DPI (Aerolizertm Inhaler) in Patients With Partially Reversible COPD
Brief Title: Formoterol Via pMDI HFA-134a Propellant or DPI in Partially Reversible Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Collaborators: Vito Brusasco "Centro Dipartimentale di Fisiopatologia Respiratoria", University of Genoa, Italy (Co-ordinating centre) (Unknown); Giovanni Barisione "Unità Operativa di Medicina Preventiva e del Lavoro, Laboratorio di Fisiopatologia Respiratoria", S. Martino Hospital, Genoa, Italy (Unknown); Universita degli Studi di Genova (Other); Cardarelli Hospital (Other); Roberto Dal Negro "Unità Operativa di Pneumologia", Hospital of Bussolengo (Verona), Italy (Unknown); University of Modena and Reggio Emilia (Other); Carlo Mereu "Struttura complessa di Pneumologia", S. Corona Hospital, Pietra Ligure (Savona), Italy (Unknown); University of Pisa (Other); Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Guido Varoli, Clinical Project Manager, Chiesi Farmaceutici S.p.A.
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DM PR 3301 002 03
Record Dates: First submitted 2008-08-26; First posted 2008-08-27 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Active Comparator): Formoterol pMDI
  Interventions: Drug: Formoterol; Drug: Placebo
- B (Active Comparator): Formoterol dry powder
  Interventions: Drug: Formoterol; Drug: Placebo
- C (Placebo Comparator): Placebo pMDI DPI
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Formoterol — pMDI 12 mcg/dose 1 dose in the morning and 1 dose in the evening
  Other Names: Atimos
  Arms: A
Drug: Formoterol — DPI 12 mcg/dose 1 dose in the morning and 1 dose in the evening
  Other Names: Foradil
  Arms: A; B
Drug: Placebo — Placebo pMDI/DPI 1 dose in the morning and 1 dose in the evening

SUMMARY:
The purpose of this study is to demonstrate equivalent efficacy between two different formulations of formoterol (pMDI using HFA-134 propellant and dry powder) on lung function in adult patients with partially reversible COPD.

DETAILED DESCRIPTION:
The present study is aimed at investigating the effect of a single 12 µg dose and of a short 7-day course of formoterol HFA-134a, compared to a formoterol DPI formulation, on specific parameters that are appropriate for assessment of single-dose and short-term effects on COPD.

This study has been designed to assess the efficacy with the traditional use of FEV1. Furthermore, the use of other efficacy parameters such as changes in exertion tolerance and dyspnoea, dynamic and static volumes measured using a whole body plethysmograph, such as TLC, RV, IC and airways conductance sGAW has been included.

This is a double blind, double dummy, multicentre, randomised, placebo-controlled, cross-over study in at least 36 adult patients with partially reversible COPD. The two test treatments and placebo will be administered in a single and repeated (twice daily for 7 days) dose cycle (with a minimum 2 days and maximum 7 days of wash-out between each cycle).

Seven clinic visits in total will take place at the start and end of the run-in period, and at the first and at the last dose of each treatment cycle (with placebo and the two active treatment tests), with an acceptable variation of a maximum of ± 1 day in respect of the scheduled days at the end of each treatment cycle (i.e. treatment with placebo or active drug may range between 6 and 8 days).

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex aged > 40 years.
* Clinical diagnosis of partially reversible COPD, with or without chronic symptoms, in line with the following recommendations of the National Heart Lung and Blood Institute/World Health Organisation (NHLBI/WHO) Global Initiative for Chronic Obstructive Lung Disease (GOLD) (22):
* Post-bronchodilator FEV1 ≥ 30% and < 80% of the predicted normal values, and at least 0.7 L (if less than 0.7 L, FEV1 must be ≥ 40% of predicted normal value)
* FEV1/FVC ratio < 70%.
* Positive partial response to the reversibility test in the screening visit, defined as an increase from baseline value of at least 5% of the percentage of predicted normal value (post-dosing minus pre-dosing/pre-dosing x 100) in the FEV1 measurement 30 minutes following 4 puffs (4 x 100 µg) of inhaled salbutamol pMDI.
* Current or past tobacco heavy smoking habits (defined as smoking for > 20 pack years, where 1 pack year = 20 cigarettes/day for 1 year or equivalent).
* A cooperative attitude and ability to be trained to use correctly the pMDI and the AerolizerTM inhaler.
* Written informed consent obtained.

Exclusion Criteria:

* Evidence of COPD exacerbation and/or symptomatic infection of the airways in the previous 4 weeks requiring antibiotic therapy.
* History of clinically significant disease whose sequelae and/or treatments can interfere with the results of the present study.
* Presence of asthma.
* Evidence of bronchiectases.
* History of inadequate cardiac, hepatic and/or renal function.
* History of coronary artery disease, myocardial infarction, cerebrovascular disease, cardiac arrhythmias, severe hypertension and diabetes mellitus.
* Other haemodynamic relevant rhythm disturbances (including atrial flutter or atrial fibrillation with ventricular response, bradycardia (≤ 55 bpm), evidence of atrial-ventricular (AV) block on ECG of more than 1st degree.
* History of percutaneous transluminal coronary angioplasty (PTCA) or coronary artery by-pass graft (CABG).
* Patients with a serum potassium value ≤ 3.5 mEq/L and/or serum glucose value ≥ 140 mg/dL.
* Patients with an abnormal QTc interval value in the ECG test, defined as > 450 msec in males or > 470 msec in females.
* Evidence of posture and gait disturbances, or impairment of limb coordination due to any cause.
* Patients taking oral corticosteroids in the last month prior to study entry.
* Patients taking inhaled long-acting β2-agonists or anticholinergics in the last 48 hours.
* Patients already taking inhaled corticosteroids (including nasal), sodium cromoglycate and nedocromil sodium, leukotriene antagonists, xanthyne derivatives, mucolytics, antitussives for whom the dose has been changed in the last month before study entry or is likely to change during the total study period.
* History of hypersensitivity to sympathomimetic drugs.
* Patients taking β-antagonists, tricyclic antidepressants or monoamine oxidase inhibitors (MAOI).
* Pregnant or lactating females or females at risk of pregnancy, i.e. those not demonstrating adequate contraception (i.e. barrier methods, intrauterine devices, hormonal treatment or sterilization). A pregnancy test is recommended - Patients with a post-bronchodilator FEV1 < 0.7 L and with a predicted normal FEV1 < 40%.
* Patients requiring long-term oxygen therapy.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2004-09; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
FEV1 area under the curve (AUC) standardized for time | 4 hours following the morning dose of study medication at the first visit of each treatment cycle

SECONDARY OUTCOMES:
Clinical equivalence in terms of FEV1 area under the curve (AUC) standardized for time | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Barisione, MD, Principal Investigator — "Unità Operativa di Medicina Preventiva e del Lavoro, Laboratorio di Fisiopatologia Respiratoria", S. Martino Hospital, Genoa, Italy; Giorgio Canonica, MD, Principal Investigator — 3) "Clinica di Malattie dell'Apparato Respiratorio e Allergologia, Dipartimento di Medicina Interna", University of Genoa, Italy; Gennaro D'Amato, MD, Principal Investigator — 'Unita' di Pneumologia e Allergologia, Dipartimento di Medicina Respiratoria', A. Cardarelli Hospital, Naples, Italy; Roberto Dal Negro, MD, Principal Investigator — 5) "Unità Operativa di Pneumologia", Hospital of Bussolengo (Verona), Italy; Leonardo Fabbri, MD, Principal Investigator — "Clinica di Malattie dell'Apparato Respiratorio", University of Modena, Italy; Carlo Mereu, MD, Principal Investigator — "Struttura complessa di Pneumologia", S. Corona Hospital, Pietra Ligure (Savona), Italy; Pierluigi Paggiaro, MD, Principal Investigator — "Servizio di Fisiopatologia Respiratoria, Dipartimento Cardiotoracico", University of Pisa, Italy; Giorgio Scano, MD, Principal Investigator — "Unità Operativa di Riabilitazione Respiratoria, Fondazione Don Carlo Gnocchi ONLUS", Pozzolatico (FI), Italy; Vito Brusasco, MD, PhD, Study Director — "Centro Dipartimentale di Fisiopatologia Respiratoria", University of Genoa, Italy (Co-ordinating centre)
Locations (1):
- "Centro Dipartimentale di Fisiopatologia Respiratoria", University of Genoa, Genova, Italy

REFERENCES:
- [Result] Brusasco V, Canonica GW, Dal Negro R, Scano G, Paggiaro P, Fabbri LM, Barisione G, D'Amato G, Varoli G, Baroffio M, Milanese M, Mereu C, Crimi E. Formoterol by pressurized metered-dose aerosol or dry powder on airway obstruction and lung hyperinflation in partially reversible COPD. J Aerosol Med Pulm Drug Deliv. 2011 Oct;24(5):235-43. doi: 10.1089/jamp.2010.0862. Epub 2011 Jun 20. PMID 21689019